CLINICAL TRIAL: NCT02982070
Title: TU (University of Tulsa) Tough: Mental Toughness Training for College Success
Brief Title: TU Tough: Mental Toughness Training for College Success
Acronym: TUtough
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016-004
Record Dates: First submitted 2016-11-29; First posted 2016-12-05 (Estimated); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Stress, Psychological
Keywords: psychological well-being, academic success
MeSH Terms: conditions — Stress, Psychological; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mental Toughness Training (Experimental): Behavioral training in goal-building, mindfulness, and the growth mindset.
  Interventions: Behavioral: Mental Toughness Training
- College as Usual (No Intervention): no training provided

INTERVENTIONS:
Behavioral: Mental Toughness Training — Behavioral training in goal-building, mindfulness, and the growth mindset.
  Other Names: Resiliency training
  Arms: Mental Toughness Training

SUMMARY:
The aims of this study are to (1) assess the extent of psychological distress for incoming first-year students at the University of Tulsa (Part 1), (2) assess the impact of "mental toughness" training on the trajectory of psychological well-being and academic success (Part 2), (3) assess the impact of mental toughness training on neural and behavioral reactivity to affective stimuli and decisions (Part 3), and (4) examine genetic markers of resiliency in college populations and interactions between genetic markers and response to mental toughness training (Part 2).

DETAILED DESCRIPTION:
Part 1 will consist of an online survey, sent by email. This email will be sent through the TU (University of Tulsa) Student Affairs office to all incoming freshman students and will also be sent by study personnel to students who indicate interest in the study through the other recruitment efforts (i.e., flyers on campus). This survey will also allow students to indicate whether or not they would be interested in being involved in future research regarding mental toughness and strategies for college success. The second aim will be accomplished via Part 2 of the study. Part 2 is the longitudinal portion that assesses students' well-being (i.e., happiness, distress, anxiety, satisfaction, etc.) and academic success (i.e., retention at TU, GPA, etc.) before and after completion of either mental toughness training or "college as usual". These participants will be selected from the group of participants who complete Part 1 and/or via ongoing courses within each college at the university (see recruitment section). Part 2 will enroll a maximum of 300 participants/year for the first 3 years, each of whom will then be asked to remain in the study for 5 years. These participants will be contacted via phone, text message, or email to determine whether they are interested and meet criteria. Those who meet criteria will be scheduled for an in-person session at TU (Part 2) to complete written informed consent, provide the saliva sample, obtain instructions regarding the completion of survey sessions and the training protocol. Those who enroll in this study will then be asked to complete survey sessions repeatedly over the next 5 years: (1) During the first semester, Part 2 participants will be asked to complete three survey sessions, one pre- and one post- training phase, and one during finals week. (2) During the Spring semester of the first year, each participant would complete three surveys (within the first two weeks; mid semester; and during finals week), followed by one survey mid-Summer. (3) For Years 2-5, survey sessions would occur once per semester (Fall, Spring, Summer), allowing examination of how training may impact longer-term trajectories of academic success and psychological well-being. Each online surveys will assess for psychological well-being, demographics and medical history, and academic activities. For those who provide consent for us to access limited information from academic records (as specified in the consent and in the research protocol section of this document), the information will be combined with the collected survey data. For Part 3, data will be collected from a subset of participants during two neuroimaging sessions at LIBR (Laureate Institute for Brain Research). The first neuroimaging session will be completed within one month of beginning the training phase (mental toughness or "college as usual") and the second will be completed within one month of the end of the training phase. Each neuroimaging session will last approximately 3-4 hours and will involve completion of self-report measures regarding current affective state, a behavioral measure of exploratory behavior, and a functional MRI session during which participants will complete tasks related to processing of emotional faces, emotional images, and reward. The fourth aim will also be accomplished via Part 2 of the study, which involves the collection of DNA saliva collection once during the first semester of their first year. Samples will be collected in-person at their first baseline session, after written informed consent is obtained. This data will be used to assess any genetic markers of resiliency that exist in college populations and to determine if there are genetic markers that interact with the impact of mental toughness training (i.e., if individuals with specific genetic markers do better or worse with training).

ELIGIBILITY:
Inclusion Criteria:

1. Age: 17 years old and over as of the first day of classes at TU for the year they are being enrolled in the study. Due to this, all participants will be 18 years of age or older when completing Year 2 of the longitudinal aspect of the study (Part 2, Component B and C). A separate section concerning the inclusion of minors has been included below.
2. Are an incoming first year student at the University of Tulsa
3. All genders
4. All races
5. Able to provide informed consent (or, if 17, to have their parents complete informed consent and the minor complete informed assent).
6. Have sufficient proficiency in English language to understand and complete interviews, questionnaires, and all other study procedures.
7. Have regular access to a personal, campus, or other computer on which to complete online surveys.
8. For Part 3 only (neuroimaging portion), participants must have at least normative levels of perceived stress (>21), as determined by the mean score from the initial survey session completed under protocol 2015-010. This is to identify participants who have the greatest potential to show demonstrable symptomatic change with mental toughness training.

Exclusion Criteria (for Part 3, neuroimaging portion only):

1. Has a history of unstable liver or renal insufficiency; glaucoma; significant and unstable cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, or metabolic disturbance; or any other condition that, in the opinion of the investigator, would make participation not be in the best interest (e.g., compromise the well-being) of the subject or that could prevent, limit, or confound the protocol-specified assessments.
2. Current use of a medication that could potentially affect brain functioning (e.g., stimulants, antidepressants, anxiolytics, antipsychotics, mood stabilizers, anti-hypertensives). Inclusion of individuals reporting other types of medications or supplements not listed or considered thus far will be at the discretion of the PI according to evidence in the literature of it affecting brain function or brain blood flow.
3. MRI contraindications including: cardiac pacemaker, metal fragments in eyes/skin/body (shrapnel), aortic/aneurysm clips, prosthesis, by-pass surgery/coronary artery clips, hearing aid, heart valve replacement, shunt (ventricular or spinal), electrodes, metal plates/pins/screws/wires, or neuro/bio-stimulators (TENS unit), persons who have ever been a professional metal worker/welder, history of eye surgery/eyes washed out because of metal, vision problems uncorrectable with lenses, inability to lie still on one's back for 60-120 minutes; prior neurosurgery; tattoos or cosmetic makeup with metal dyes, unwillingness to remove body piercings, and pregnancy.
4. Moderate to severe traumatic brain injury (>30 min. loss of consciousness or >24 hours posttraumatic amnesia) or other neurocognitive disorder with evidence of neurological deficits, neurological disorders, or severe or unstable medical conditions that might be compromised by participation in the study (to be determined by primary care provider)
5. Non-correctable vision or hearing problems

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 538 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2023-03-18 (Actual); Study Completion 2023-07-23 (Actual)

PRIMARY OUTCOMES:
Grade point average (GPA) | Last semester that students are enrolled at the university, on average after 3.5 years.
  GPA obtained from academic records
Retention in college | Last semester that students are enrolled at the university, on average after 3.5 years.
  Retention assessed as whether or not the student remains enrolled in the university.
Change in Connor---Davidson Resilience Scale (CD---RISC 10) | Baseline and completion of training, on average after 4 weeks.
  This measure assessed characteristics associated with resiliency and mental toughness.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Scale | Baseline and completion of training, on average after 4 weeks.
  This measure assesses symptoms of anxiety over the past 7 days.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Scale | Baseline and completion of training, on average after 4 weeks.
  This measure assesses symptoms of depression.

SECONDARY OUTCOMES:
National Institute of Health Toolbox Perceived Stress Scale | Average across all time points from post-training (average of 4 weeks after baseline) to the last semester they are enrolled at the university, (on average 3.5 years after baseline).
  This measure assesses the level of stress experienced over the past month.
Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Scale | Average across all time points from post-training (average of 4 weeks after baseline) to the last semester they are enrolled at the university, (on average 3.5 years after baseline).
  This measure assesses symptoms of anxiety over the past 7 days.
Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Scale | Average across all time points from post-training (average of 4 weeks after baseline) to the last semester they are enrolled at the university, (on average 3.5 years after baseline).
  This measure assesses symptoms of depression over the past 7 days.
Change in percent signal change within anatomically-defined medial prefrontal cortex, amygdala, dorsolateral prefrontal cortex, anterior insula, and ventral striatum. | Baseline and completion of training, on average after 4 weeks.
  Change in percent signal change within anatomically-defined medial prefrontal cortex and amygdala (during emotional face processing), dorsolateral prefrontal cortex and anterior insula (during decision-making), and ventral striatum (during reward processing).
Resting state connectivity between brain regions | Baseline and completion of training, on average after 4 weeks.
  Resting state connectivity between brain regions

CONTACTS AND LOCATIONS:
Overall Officials: Robin Aupperle, PhD, Principal Investigator — Laureate Institute for Brain Research
Locations (2):
- United States (2):
  - The University of Tulsa, Tulsa, Oklahoma
  - Laureate Institute for Brain Research, Tulsa, Oklahoma

IPD SHARING:
Plan to Share IPD: No